CLINICAL TRIAL: NCT04112251
Title: Effect of Cocoa Flavonols Oral Supplement on Body Composition, Metabolic, Inflammatory and Oxidative Profile in Obese Subject 10 to 16 Years
Brief Title: Effects of COcoa Supplement in OBese Adolescent Subjects
Acronym: COOBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Polytechnic Institute, Mexico (Other)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Instituto Nacional de Salud Publica, Mexico (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Guillermo Ceballos Reyes, Researcher, National Polytechnic Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COOBA-HIM-100
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Childhood Obesity; Adolescent Obesity
Keywords: Childhood Obesity; Cocoa Flavanols; Adolescent Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Catechin

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical trial will be conducted, which will be conducted at the Federico Gómez Children's Hospital in Mexico, during the period from October 2019 to October 2020; with patients with exogenous obesity from 10 to 16 years.
Who Masked: Participant, Care Provider, Investigator
Masking Description: For the implementation of the intervention, they are masked by means of the following measures:
  1. The organoleptic characteristics of the interventions will be the same in color, smell, taste, texture, consistency, weight and size.
  2. The primary container will be the same size, and will contain 65 capsules, which will be identified by means of a code.
  3. The delivery of the treatment will be carried out by a collaborator who is not directly related to the research project, which will be assigned by the Hospital's clinical epidemiology area, according to the randomization list sent by the Integral Cardiometabolic Research Laboratory of the Polytechnic Institute National, in a sealed security envelope.
  4. No direct participant should adjust the dose of the treatment, during the follow-up they will only verify the attachment of the intervention based on the capsule count, collection of anecdotes and direct interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This group will receive the usual therapy of the endocrinology service, dietary recommendations, physical activity recommendations and the administration of a 500 mg oral placebo capsule (Cornstarch) every 12 hours for 12 weeks.
  Interventions: Dietary Supplement: Cocoa Flavonols Supplement
- Supplement (Experimental): This group will receive the usual therapy of the endocrinology service, dietary recommendations, physical activity recommendations and the administration of a 500 mg capsule every 12 hours (100 mg / day of epicatechin) for 12 weeks.
  Interventions: Dietary Supplement: Cocoa Flavonols Supplement

INTERVENTIONS:
Dietary Supplement: Cocoa Flavonols Supplement — Whose total capsule content of 500 mg of cocoa flavonoids, 50 mg correspond to (-) - epicatechin per capsule, with a total dose of this compound being 100 mg/day.
  Other Names: (-)-epicatechin

SUMMARY:
Childhood obesity is a serious public health problem internationally. In addition to being associated with the early onset of chronic degenerative diseases such as diabetes, dyslipidemias, coronary artery diseases, among others.

Changes in lifestyle habits are the main axis in the treatment of this disease; however, low adherence to these changes are reflected in the increase in their incidence and prevalence.

There is diverse evidence that the use of flavonoids from cocoa such as (-) - epicatechin are able to prevent cardiovascular risks, decrease insulin resistance, mean arterial pressure, control the lipid profile; mediate oxidative stress, improve mitochondrial function and regulate the inflammatory process in patients with heart failure and diabetes mellitus. Therefore, our working hypothesis is the administration of the oral supplement of flavonoids from cocoa for 12 weeks will be able to reduce the percentage of body fat, improve the metabolic profile and regulate inflammatory and oxidative processes in obese patients 10-16 years, compared to those patients who only take a usual therapy consisting of recommendations of healthy diet and physical activity.

For this, a randomized, double-blind, placebo-controlled clinical trial will be carried out, which will be carried out at the Federico Gómez Children's Hospital of Mexico, during the period from October 2019 to October 2020; with obese patients from 10 to 16 years distributed homogeneously at random in two groups: the control group (Placebo) and the intervention group (Flavonoids from cocoa) both groups affected for 12 weeks.

The variables studied will be: percentage of muscle mass, percentage of fat, body mass index (BMI), waist circumference (CC), fasting glucose, fasting insulin, lipid profile (Total cholesterol, Triglycerides, HDL-c, LDL -c, Ratio TG / HDL-c, High Sensitivity C-Reactive Protein (HS-CRP), Interleukins (IL-6, IL-10), Tumor Growth Factor beta (TGF-β) and Tumoral Necrosis Factor alpha (TNF-α), carbonylated proteins, Malondialdehyde (MDA), indirect calorimetry by respiratory coefficient and treatment adherence.

DETAILED DESCRIPTION:
Childhood obesity is global health problem, due to the constant increase in its incidence and prevalence. Having this disease helps increase the costs of care for Chronic Noncommunicable Diseases. The increase in its prevalence since 1975 from 1% to 6% (girls) and 8% (boys) in 2016 between the ranges of 5 to 19 years.

Mexico, occupies the first place worldwide in childhood obesity, only by data from National Health and Nutrition Survey 2016 , it is considered that approximately 3 out of 10 children, 4 out of 10 adolescents present this health problem; the population with the highest health risk being ages between 10 and 17 years. In 2016, the prevalence of obesity in the population between 5 and 11 years old was 15.3% and in adolescents between 12 and 19 years old it was 13.9% .

Although, the scientific evidence has focused on studying different strategies for the prevention, control and treatment of childhood obesity complications; The prevalence of this has not yet been reduced or controlled favorably. It has been demonstrated through meta-analysis and randomized clinical trials that the use of flavonoids from cocoa, such as epicatechin at a concentration of 50 mg to 100 mg / day for 6 to 18 weeks, may decrease the risk of cardiovascular and metabolic diseases, Because it reduces: insulin resistance, diastolic blood pressure, triglycerides, LDL-c and increased HDL-c. These biological effects are related to the antioxidant capacity (inhibition of Nicotinamide adenine dinucleotide phosphate oxidase (NAHPH) and increase of endothelial Nitric Oxide Synthase (eNOS), protein interaction and cell signaling that these compounds have (inhibition of Tumoral Necrosis Factor alpha (TNF-α) and Necrosis Factor beta (NF-β); MAPK pathway regulation ) and finally by the regulation of the inflammatory process through the modulation of the pro-inflammatory elements (Decrease of Il-6, TNF-α and PCR-HS), so it is attractive to establish it as an alternative treatment to reduce the risk of generate comorbidities This research aims to solve the following question: What is the effect of oral supplementation of flavonoids from cocoa on body composition, metabolic, inflammatory and oxidative profile in obese patients 10-16 years old?

This work aims to demonstrate the effect of oral supplementation of flavonoids from cocoa on body composition, anthropometric parameters, biochemical, inflammatory and oxidative markers in obese patients in order to reduce the risk of suffering from other comorbidities, such as metabolic syndrome. , diabetes, high blood pressure and cardiovascular diseases.

From this study the investigators can know the effectiveness of the use of flavonoids from cocoa as epicatechin in a child population and demonstrate the regulatory effect of epicatechin on lipids, inflammation and oxidation. The results obtained from this research will provide us with the necessary evidence to propose whether the use of these flavonoids to prevent the occurrence of other comorbidities of childhood obesity.

Material and methods:

Type of study and universe: A randomized, double-blind, placebo-controlled clinical trial will be conducted, which will be conducted at the Federico Gómez Children's Hospital in Mexico, during the period from October 2019 to October 2020; with patients with exogenous obesity from 10 to 16 years.

Sample size:

It was calculated by the G * Power software version 3.1, considering an alpha error of 0.05, a power of 95% and a minimum expected difference between groups: control and intervention based on the variables of interest according to the reports of Other studies. Assuming that the sample size with the largest number of subjects (n = 40 subjects) is sufficient to find significant differences in all the variables of interest. Once the minimum necessary sample size (40 subjects per group) for the research protocol has been calculated, the sample adjustment for losses of 30% will be made, with a total of 116 research subjects (58 for each group).

Description of the intervention:

Phase 1. Generation of healthy habits: In order to standardize patients to establish greater control in the recommendations of diet and physical activity, the implementation of educational workshops 4 weeks before the start of the intervention was considered. The content of the recommendations workshops for a healthy diet and physical activity is based on the recommendations issued by World Health Organization (WHO), Official Mexican Standard of the Ministry of Health (NOM-043-SSA2-2012) and the Guidelines for diabetes prevention programs.

Phase 2. Evaluation of the intervention: Once the phase of standardization of healthy habits is finished, the evaluation of the intervention will begin after the randomization of the study population, in 2 groups: Control Group (Placebo) that will receive the usual therapy of the endocrinology service, dietary recommendations, physical activity recommendations and the administration of one oral capsule of the placebo every 12 hours for 12 weeks and the Experimental group (Supplement of flavonoids from cocoa the participants will receive the usual therapy of the endocrinology service, dietary recommendations, physical activity recommendations and the administration of one capsule every 12 hours for 12 weeks.

Randomization of the sample:

For the selection of intervention and control groups, select a randomized selection of research subjects through the online Research Randomizer (www.randomizer.org) taking into account 2 unique sets, with 60 numbers per-set, a range between 1 and 120.

Blinding of the intervention:

For this study, a double blinding was established and masking techniques will be established to avoid the identification of the intervention. Blinding will only be opened when required by the research ethics committee or secretary of health, or when the patient presents a serious adverse event; same that will be informed before the competent authorities.

This work will be guided by the ethical principles for research in humans of the Helsinki Declaration 2013 and the recommendations postulated in the guide of good clinical practices issued by the WHO. In accordance with the provisions of the Regulations of the General Law on Research Health in Article 17, it is classified as a risk greater than the minimum. Currently, it has the approval of the Biosafety Committees, the Research and Research Ethics Committees of the Federico Gómez Children's Hospital of Mexico (HIM-2018-100).

Statistical analysis plan:

The data obtained from the results of this research will be subjected to an analysis by protocol and by intention to be treated. For the statistical analysis of the results, the Statistical Package for the Social Sciences Softaware by International Business Machines (IBM SPSS) version 24 program will be used. Reporting the mean and standard deviation for the quantitative variables; median and range for qualitative variables. The distribution of the sample studied will be carried out the normality test of Kolmogórov-Smirnov. For the evaluation of the changes of the variables of interest, in case of presenting a normal distribution, repeated measures ANOVA and T Student will be used for related samples. In case of presenting a free distribution will be used will be the Kruskal - Wallis and Wilcoxon tests. Finally, to evaluate the presence of changes between the groups through the covariance analysis of the deltas of change of the variables studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients 10 to 16 years old.
* Patients who do not take any pharmacological treatment for chronic conditions.
* Have the signed informed consent and assent.
* Only the participation of one research subject per family will be accepted.

Exclusion Criteria:

* Carrying diseases that can alter body weight (endocrine, hematological, immunological, neurological, psychiatric, genetic alterations).
* Presence of mental retardation and other chronic diseases.
* That they receive medications that can affect weight, lipid and carbohydrate metabolism.
* That you are actively participating in some other research protocol.
* Do not have a body limb.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
TG / HDL-C ratio | 3 month
  The Triglycerides / High-density lipoprotein cholesterol (TG / HDL-c) index is the most practical atherogenic marker for assessing the presence of cardiometabolic risks.
Body Fat Mass (BFM) percentage | 3 month
  Result obtained by dual x-ray absorptiometry
Insulin Resistance Homeostasis Evaluation Model (HOMA-IR) | 3 month
  Result obtained from fasting glucose determinations multiplied by fasting insulin determination divided by a constant of 405

SECONDARY OUTCOMES:
Quantitative determination of HS-PCR, TNF-α, TFG-β, IL-6 and IL-10 | 3 month
  Result obtained from the quantification by Kits of human inflammatory cytokines by Enzyme Linked Inmuno Sorbent Assay from blood serum.
Determined by the quantification of carbonylated protein | 3 month
  Result obtained from the quantification of absorbance by colorimetry of carbonyl groups of proteins are generated by oxidation of several chains of amino acids, by the adduct formation of the reaction of Michael and glycosylation
Determined by the quantification of Malondialdehyde (MDA) | 3 month
  Result obtained from the quantification of the absorbance by colorimetry of the decomposition of unsaturated lipids that react by the addition from Michael.
Body Mass Index (BMI) | 1 Month
  Result obtained from the division body weight and square size
Indirect Calorimetry | 3 month
  Determined by calculating the respiratory coefficient by measuring the Carbon Dioxide (CO2) produced with respect to the Oxygen (O2) consumed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aceves-Martins M, Llaurado E, Tarro L, Sola R, Giralt M. Obesity-promoting factors in Mexican children and adolescents: challenges and opportunities. Glob Health Action. 2016 Jan 18;9:29625. doi: 10.3402/gha.v9.29625. eCollection 2016. PMID 26787421
- [Result] Grant-Guimaraes J, Feinstein R, Laber E, Kosoy J. Childhood Overweight and Obesity. Gastroenterol Clin North Am. 2016 Dec;45(4):715-728. doi: 10.1016/j.gtc.2016.07.007. PMID 27837784
- [Result] Kim J, Lee I, Lim S. Overweight or obesity in children aged 0 to 6 and the risk of adult metabolic syndrome: A systematic review and meta-analysis. J Clin Nurs. 2017 Dec;26(23-24):3869-3880. doi: 10.1111/jocn.13802. Epub 2017 May 23. PMID 28295797
- [Result] Gupta N, Goel K, Shah P, Misra A. Childhood obesity in developing countries: epidemiology, determinants, and prevention. Endocr Rev. 2012 Feb;33(1):48-70. doi: 10.1210/er.2010-0028. Epub 2012 Jan 12. PMID 22240243
- [Result] Peneau S, Giudici KV, Gusto G, Goxe D, Lantieri O, Hercberg S, Rolland-Cachera MF. Growth Trajectories of Body Mass Index during Childhood: Associated Factors and Health Outcome at Adulthood. J Pediatr. 2017 Jul;186:64-71.e1. doi: 10.1016/j.jpeds.2017.02.010. Epub 2017 Mar 7. PMID 28283258
- [Result] Zlatohlavek L, Hubacek JA, Vrablik M, Pejsova H, Lanska V, Ceska R. The Impact of Physical Activity and Dietary Measures on the Biochemical and Anthropometric Parameters in Obese Children. Is There Any Genetic Predisposition? Cent Eur J Public Health. 2015 Nov;23 Suppl:S62-6. doi: 10.21101/cejph.a4191. PMID 26849546
- [Result] Marseglia L, Manti S, D'Angelo G, Nicotera A, Parisi E, Di Rosa G, Gitto E, Arrigo T. Oxidative stress in obesity: a critical component in human diseases. Int J Mol Sci. 2014 Dec 26;16(1):378-400. doi: 10.3390/ijms16010378. PMID 25548896
- [Result] Faienza MF, Francavilla R, Goffredo R, Ventura A, Marzano F, Panzarino G, Marinelli G, Cavallo L, Di Bitonto G. Oxidative stress in obesity and metabolic syndrome in children and adolescents. Horm Res Paediatr. 2012;78(3):158-64. doi: 10.1159/000342642. Epub 2012 Oct 10. PMID 23052543
- [Result] Becker K, Geisler S, Ueberall F, Fuchs D, Gostner JM. Immunomodulatory properties of cacao extracts - potential consequences for medical applications. Front Pharmacol. 2013 Dec 12;4:154. doi: 10.3389/fphar.2013.00154. PMID 24376420
- [Result] Almoosawi S, Tsang C, Ostertag LM, Fyfe L, Al-Dujaili EA. Differential effect of polyphenol-rich dark chocolate on biomarkers of glucose metabolism and cardiovascular risk factors in healthy, overweight and obese subjects: a randomized clinical trial. Food Funct. 2012 Oct;3(10):1035-43. doi: 10.1039/c2fo30060e. Epub 2012 Jul 16. PMID 22796902
- [Result] Gutierrez-Salmean G, Ortiz-Vilchis P, Vacaseydel CM, Rubio-Gayosso I, Meaney E, Villarreal F, Ramirez-Sanchez I, Ceballos G. Acute effects of an oral supplement of (-)-epicatechin on postprandial fat and carbohydrate metabolism in normal and overweight subjects. Food Funct. 2014 Mar;5(3):521-7. doi: 10.1039/c3fo60416k. PMID 24458104
- [Result] Gutierrez-Salmean G, Meaney E, Lanaspa MA, Cicerchi C, Johnson RJ, Dugar S, Taub P, Ramirez-Sanchez I, Villarreal F, Schreiner G, Ceballos G. A randomized, placebo-controlled, double-blind study on the effects of (-)-epicatechin on the triglyceride/HDLc ratio and cardiometabolic profile of subjects with hypertriglyceridemia: Unique in vitro effects. Int J Cardiol. 2016 Nov 15;223:500-506. doi: 10.1016/j.ijcard.2016.08.158. Epub 2016 Aug 8. PMID 27552564
- [Result] Al-Khudairy L, Loveman E, Colquitt JL, Mead E, Johnson RE, Fraser H, Olajide J, Murphy M, Velho RM, O'Malley C, Azevedo LB, Ells LJ, Metzendorf MI, Rees K. Diet, physical activity and behavioural interventions for the treatment of overweight or obese adolescents aged 12 to 17 years. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012691. doi: 10.1002/14651858.CD012691. PMID 28639320
- [Result] Mead E, Brown T, Rees K, Azevedo LB, Whittaker V, Jones D, Olajide J, Mainardi GM, Corpeleijn E, O'Malley C, Beardsmore E, Al-Khudairy L, Baur L, Metzendorf MI, Demaio A, Ells LJ. Diet, physical activity and behavioural interventions for the treatment of overweight or obese children from the age of 6 to 11 years. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012651. doi: 10.1002/14651858.CD012651. PMID 28639319
- See also: Worldwide epidemiological data of childhood obesity — http://www.who.int/mediacentre/news/releases/2017/increase-childhood-obesity/es/.
- See also: Epidemiological data of childhood obesity in Mexico — https://www.gob.mx/cms/uploads/attachment/file/209093/ENSANUT.pdf
- See also: Beneficial effects of a flavanol-enriched cacao beverage on anthropometric and cardiometabolic risk profile in overweight subjects — https://www.medigraphic.com/cgi-bin/new/resumenI.cgi?IDARTICULO=58908